CLINICAL TRIAL: NCT04927234
Title: Postoperative Oedema Management of Foot and Ankle Patients With Neuromuscular Electro-stimulation of the Peroneal Nerve Using Geko™
Brief Title: Foot and Ankle Post-operative Oedema Management Using Geko™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firstkind Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FSK-F&A-001
Record Dates: First submitted 2021-06-03; First posted 2021-06-15 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Surgery; Edema
Keywords: geko; foot surgery; ankle surgery; oedema management; post-operative oedema
MeSH Terms: conditions — Edema

STUDY DESIGN:
Intervention Model Description: Standard block randomisation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of care + geko™ Therapy (Experimental): In addition to their standard of care, for patients randomised to the intervention arm, geko™ therapy will be applied immediately post-surgery on the operated leg and administered for 24 hours / day whilst the patient remains in hospital, after which geko™ therapy will then be applied for 12hrs / day until the patient returns for their first post-operative follow-up visit (Day 14 ± 2 days post-surgery)
  Interventions: Device: geko™ therapy
- Standard of care (No Intervention): Patients will receive their standard of care as per hospital practice.

INTERVENTIONS:
Device: geko™ therapy — Neuro-muscular electrical stimulation of the peroneal nerve
  Other Names: geko; NMES
  Arms: Standard of care + geko™ Therapy

SUMMARY:
The multicentre randomised geko™ Foot and Ankle Trial will prospectively and systematically collect clinical data on patients randomised, on a 1:1 basis, to either standard care or standard care plus geko™ therapy to assess oedema management and patient outcomes during a follow-up period of up to three months post-surgery.

DETAILED DESCRIPTION:
The geko™ device has a wide range of clinical applications including the post-operative management of oedema.

Although many short-term acute studies have been completed using the device, little clinical data has been collected on the effect of geko™ use in current standard care pathways for oedema management on patient outcomes during long term follow-up after surgery.

This study is an open label, multi-centre prospective randomised study. The study patient population will be randomised on a 1:1 basis into two groups of 61 patients each. These groups are defined as Group A patients who receive geko™ therapy and SC i.e. the intervention group and Group B patients who receive Standard Care (SC) only i.e. no intervention. The participants will be assessed pre-surgery and up to 90 days post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years
* Intact healthy skin at the site of geko™ device application.
* Patients that have been listed for forefoot and / or hindfoot surgery
* Patient understands and is willing to participate in the study and can comply with study procedures
* Patient is willing and able to give written informed consent

Exclusion Criteria:

* Pregnant
* Use of any other neuro-modulation device.
* Trauma to the lower limbs that would prevent geko™ from stimulating the common peroneal nerve.
* No response to geko™ therapy i.e. no involuntary rhythmic upward and outward movement of the foot (dorsiflexion) at the maximum tolerable device setting
* Participation in any other clinical study that may interfere with the outcome of either study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-08-05 (Actual)

PRIMARY OUTCOMES:
Assessment of post-operative oedema formation using the figure-of-eight tape measurement | From pre-surgery assessment until up to 90 days post-surgery
  To assess the effect of geko™ therapy on oedema formation following foot and / or ankle surgery. This will be done using the figure of eight tape measurement method
Assessment of post-operative oedema formation using the pitting oedema scale | From pre-surgery assessment until up to 90 days post-surgery
  To assess the effect of geko™ therapy on oedema formation following foot and / or ankle surgery using the pitting oedema scale, where following a 2 second firm thumb press, 0 (min) indicates no oedema and 4 (max) is a very deep pit.
Assessment of post-operative oedema formation using bioimpedance analysis (US sites only) | From pre-surgery assessment until up to 90 days post-surgery
  To assess the effect of geko™ therapy on oedema formation following foot and / or ankle surgery using a bioimpedance device to measure resistance to electrical current in both legs and calculating the percentage difference between the operated leg and the contralateral limb.

SECONDARY OUTCOMES:
Incidence of Adverse Events in each group | From pre-surgery assessment until up to 90 days post-surgery
Incidence of device deficiencies | from start of geko treatment (immediately post-surgery) until up to 90 days post-surgery
  To assess the number of geko device deficiencies (if any)
Change in pain level using a visual analogue scale (VAS) score | From pre-surgery assessment until up to 90 days post-surgery
  Assessing pain levels using a visual analogue scale (VAS) score, where 0 means no pain and 100 is the worst pain possible.
Incidence of surgical wound healing | From surgery until up to 90 days post-surgery
  Visually assessing the surgical wound healing status as either healed/progressing/static/deteriorating/severe.
Change in analgesia dosage | From pre-surgery assessment until up to 90 days post-surgery
  Assessing changes in dosage of recorded analgesic medication taken by the patient
Change in analgesia frequency | From pre-surgery assessment until up to 90 days post-surgery
  Assessing changes of frequency of recorded analgesic medication taken by the patient
Change in patient reported outcomes via Manchester-Oxford Foot & Ankle Questionnaire (MOxFQ) | From pre-surgery assessment until up to 90 days post-surgery
  Domains that are assessed in this questionnaire include walking/standing, pain and social interaction. Scores will range from 0 to 100, where 100 is most severe.

CONTACTS AND LOCATIONS:
Overall Officials: Shelain Patel, MB BS BSc(Hons) FRCS, Principal Investigator — Royal National Orthopaedic Hospital
Locations (5):
- Golden State Orthopedics and Spine, Capitola, California, United States
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
- United Kingdom (2):
  - Maidstone and Tunbridge Wells NHS Trust, Royal Tunbridge Wells
  - The Royal National Orthopaedic Hospital NHS Trust, Stanmore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Device official website — http://www.gekodevices.com/en-uk/